CLINICAL TRIAL: NCT05542849
Title: The Efficacy and Tolerability of Acarbose in Healthy Individuals: A Prospective Trial for Acarbose in Healthy Individuals Assessing Safety and Efficacy in Reducing Glucose Spikes After Carbohydrate Consumption.
Brief Title: The Efficacy and Tolerability of Acarbose in Healthy Individuals
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AgelessRx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALRx006
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Tolerance; Side Effect; Glucose Response
MeSH Terms: interventions — Acarbose

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Acarbose Tablets 50mg
- Arm B (Experimental)
  Interventions: Drug: Acarbose Tablets 50mg

INTERVENTIONS:
Drug: Acarbose Tablets 50mg — Acarbose is an Alpha-glucosidase inhibitor. It is a compound also known under the names Glucobay, Precose, and Prandase. Acarbose is used (with diet and other medications) to treat type 2 diabetes (condition in which the body does not use
  insulin normally and therefore cannot control the amount of sugar in the blood). Acarbose works by blocking α- glucosidase, which breaks down starch (aka amylose) into glucose (sugar) into your blood. Slowing food digestion
  helps keep blood glucose from rising very high after meals.

SUMMARY:
A Prospective Trial for Acarbose in Healthy Individuals Assessing Safety and Efficacy in Reducing Glucose Spikes After Carbohydrate Consumption.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. Any sex
3. Any ethnicity
4. Interest in taking Acarbose off-label
5. Approved by the AgelessRx Medical team to take Acarbose
6. Willing and technically able to use and operate a CGM
7. Own a CGM-compatible phone
8. Relatively good health with only well-managed chronic diseases (hypertension, coronary artery disease, type II diabetes, etc.) clinically stable
9. Adequate cognitive function to be able to give informed consent

Exclusion Criteria:

1. Diabetes of any type
2. Taking metformin or any other glucose lowering medication
3. Any uncontrolled endocrine disorder (thyroid, pancreatic, adrenal, etc...)
4. Active malignancy of any kind
5. Clinically relevant renal or kidney disease or dysfunction
6. History of eating disorder
7. Taking any medication, or has any medical condition that might interfere with the action of acarbose of the CGM sensor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Monophasic glucose response | 120 minutes per phase, recorded on 4 separate occasions over 2 weeks.
  Blood glucose (mg/dl) response following high carbohydrate intake

SECONDARY OUTCOMES:
Tolerability of Side Effect | Recorded on 4 separate occasions over 2 weeks.
  Tolerance of side effect profile (Scale 0 - 10) denoting no side effect at all to intolerable

CONTACTS AND LOCATIONS:
Locations (1):
- AgelessRx, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided